CLINICAL TRIAL: NCT03031314
Title: Comparison of Knotless Barbed Suture and Standard Suture in Knee Replacement Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington Hospital Healthcare System (Other)
Responsible Party: Principal Investigator, Alexander Sah, MD, Physician and Research Chair, Institute for Joint Restoration and Research, Washington Hospital Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: WHHSIJRR001
Record Dates: First submitted 2017-01-08; First posted 2017-01-25 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
Keywords: Joint Replacement; Knee Replacement; Wound Healing; Hip Replacement
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Standard suture (Active Comparator): standard suture used (monocryl)
  Interventions: Device: standard suture
- Barbed suture (Active Comparator): barbed suture used (Quill suture, Surgical Specialties)
  Interventions: Device: barbed suture

INTERVENTIONS:
Device: barbed suture
  Arms: Barbed suture
Device: standard suture
  Arms: Standard suture

SUMMARY:
Barbed suture use has been gaining increased acceptance and has been reported to offer potential advantages in wound closure of hip and knee replacement surgeries.

The goal of this study is to compare joint replacement patient outcomes who receive a knotless barbed suture versus a traditional suture (randomized into two arms). The traditional suture used at our joint replacement program is defined as: interrupted sutures to close the retinaculum followed by running monocryl sutures for skin closure. Both knotless barbed suture and the traditional sutures have similar suture size.

Patient outcomes examined will be patient range of motion (recorded daily) and complications with wound healing (evaluated periodically in-person at post-operative visits).

Secondary outcomes examined will include wound drainage on dressings by surface area and weight, as well as the wound cosmesis and perceived presence of subcutaneous surgical knots.

ELIGIBILITY:
Inclusion Criteria:

* primary joint replacement

Exclusion Criteria:

* no prior joint surgery
* no infection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Number of soft tissue infections | 12 weeks
  evaluation of wound infection after surgery, number of patients with wound infection based on clinical examination
use of antibiotics to treat infection, recorded by number | 12 weeks
  record whether antibiotics used for suspicion or treatment of superficial infection, number of episodes recorded
measurement of incision drainage, measured in grams and mm surface area | 2 weeks
  evaluation of incision drainage based on dressing saturation size and weight, measured in grams for weight, and measured by surface area mm
assessment of quality of incision closure, recorded by time and number | 12 weeks
  record delayed healing and reported by time, suture rejection based on number of episodes